CLINICAL TRIAL: NCT07200037
Title: Effects of Inspiratory Muscle Training on Weaning and Diaphragmatic Function in Prolonged Mechanical Ventilation Patients: A Multicenter Randomized Controlled Trial
Brief Title: Effects of IMT on Weaning and Diaphragmatic Function in PMV Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Shuo Chen, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250817001
Record Dates: First submitted 2025-09-02; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: Inspiratory muscle training; Prolonged mechanical ventilation; weaning

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): In this group, external load, initially 50%MIP , was daily adjusted to the highest tolerable load. The training is carried out 5 days a week for 8 weeks. The patient's MIP is measured every two weeks to adjust the training parameters in a timely manner to suit the patient's condition.
  Interventions: Behavioral: inspiratory muscle training
- sham-IMT group (Sham Comparator): In this group, external load and maximal 10% MIP remained unadjusted. The training is carried out 5 days a week. The patient's MIP is measured every two weeks to adjust the training parameters in a timely manner to suit the patient's condition.
  Interventions: Behavioral: inspiratory muscle training

INTERVENTIONS:
Behavioral: inspiratory muscle training — This intervention will include a long term program of 8 weeks IMT in PMV patients who these patients who have required at least 6h of mechanical ventilation for 21 consecutive days.

SUMMARY:
Prolonged mechanical ventilation (PMV) and weaning failure can lead to extended hospital stays, as well as increased morbidity and mortality during hospitalization. Therefore, PMV not only increases the economic burden on patients and their families, but also adds to the societal economic burden and consumes critical care medical resources. Inspiratory muscle training (IMT) is widely used by physical therapists in critically ill patients to improve respiratory function and enhance quality of life. IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function in turn promotes better respiratory function, which is clinically significant for accelerating weaning. However, most studies on the effects of IMT on weaning success rates and the duration of mechanical ventilation have limitations such as small sample sizes, homogeneous patient populations, and short intervention periods. As a result, there is still no unified, high-quality evidence-based consensus. The purpose of this study is to further clarify the role of IMT in improving diaphragmatic function and increasing weaning success rates in patients with prolonged weaning, through clinical treatment and the collection and analysis of relevant data.

DETAILED DESCRIPTION:
In recent years, inspiratory muscle training (IMT) has been widely used by physical therapists in critically ill patients to improve their respiratory function and enhance their quality of life. IMT is safe and feasible for a specific group of patients dependent on ventilators . This training not only improves inspiratory muscle strength but also increases the possibility of patients successfully being weaned off ventilators . In addition, patients who successfully weaned off the ventilator and continued with IMT also helped improve their quality of life. The current health status measured by EQ-5D VAS indicated that the symptoms of the inspiratory muscle training group improved by 12% compared with the control group. Therefore, IMT may serve as one of the training methods for physical therapists to improve the diaphragmatic function of patients with delayed weaning and increase the success rate of weaning.

In terms of the impact on the success rate of weaning from aircraft, the results of multiple randomized controlled trials and meta-analyses indicate that IMT plays a positive role in enhancing the success rate of weaning from aircraft. The results of a randomized clinical trial showed that the weaning time of the IMT group was significantly shorter than that of the control group, specifically 12.6 days compared with 18.1 days, with a P value of 0.04. This indicates that IMT can effectively shorten the duration of mechanical ventilation, thereby increasing the possibility of successful weaning. Marine pointed out in a recent article that both high-intensity IMT and low-intensity IMT can improve the MIP of patients with mechanical ventilation, increase the success rate of weaning from the ventilator and reduce the duration of mechanical ventilation, but there is no significant difference between the two groups. In addition, in this study, the forced vital capacity (FVC) of the patients increased more in the high-intensity IMT group. The absence of significant differences between the two groups in this study might be due to the fact that the study only lasted for 4 weeks, which was a relatively short intervention period. Furthermore, another systematic review revealed that although IMT could improve maximal inspiratory pressure and the Rapid Shallow Breathing Index (RSBI), no significant difference was found in the success rate of weaning from the ventilator, indicating that although IMT can enhance the strength of respiratory muscles, But it does not necessarily directly lead to a higher success rate of flight withdrawal. The effect of IMT on patients with difficult weaning due to different causes also varies. For instance, IMT studies on patients with chronic obstructive pulmonary disease (COPD) have shown that IMT not only enhances respiratory muscle strength but also improves lung function indicators, thereby improving the weaning effect. However, other studies have pointed out that the effect of IMT in patients with neuromuscular diseases is relatively limited, possibly because these patients themselves have more complex respiratory muscle weakness problems. Regarding the research on the success rate of weaning from the ventilator and the duration of mechanical ventilation by IMT, most studies have problems such as small sample size, single patient population and short intervention time. Therefore, there is no unified and high-quality evidence-based basis yet.

In conclusion, IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function will promote the improvement of respiratory function in patients, which also has certain clinical significance for accelerating weaning from the ventilator. Under the condition that our department is equipped with multiple physical therapists with experience in implementing IMT, the assessment and intervention of patients with delayed weaning in the intensive care unit were completed through the joint efforts of medical, nursing and technical staff. The success rate of weaning was the main result, and the diaphragm mobility, diaphragm thickness and diaphragm thickening fraction in the diaphragm ultrasound results were the secondary results to conduct this study. The aim is to further clarify the impact of inspiratory muscle strength training on the successful weaning of patients with delayed weaning and the improvement of diaphragmatic function through clinical treatment and data collection and analysis.

In conclusion, IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function will promote the improvement of respiratory function in patients, which also has certain clinical significance for accelerating weaning from the ventilator. Under the condition that our department is equipped with multiple physical therapists with experience in implementing IMT, the assessment and intervention of patients with delayed weaning in the intensive care unit were completed through the joint efforts of medical, nursing and technical staff. The success rate of weaning was the main result, and the diaphragm mobility, diaphragm thickness and diaphragm thickening fraction in the diaphragm ultrasound results were the secondary results to conduct this study. The aim is to further clarify the impact of inspiratory muscle strength training on the successful weaning of patients with delayed weaning and the improvement of diaphragmatic function through clinical treatment and data collection and analysis.

In conclusion, IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function will promote the improvement of respiratory function in patients, which also has certain clinical significance for accelerating weaning from the ventilator. Under the condition that our department is equipped with multiple physical therapists with experience in implementing IMT, the assessment and intervention of patients with delayed weaning in the intensive care unit were completed through the joint efforts of medical, nursing and technical staff. The success rate of weaning was the main result, and the diaphragm mobility, diaphragm thickness and diaphragm thickening fraction in the diaphragm ultrasound results were the secondary results to conduct this study. The aim is to further clarify the impact of inspiratory muscle strength training on the successful weaning of patients with delayed weaning and the improvement of diaphragmatic function through clinical treatment and data collection and analysis.

In conclusion, IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function will promote the improvement of respiratory function in patients, which also has certain clinical significance for accelerating weaning from the ventilator. Under the condition that our department is equipped with multiple physical therapists with experience in implementing IMT, the assessment and intervention of patients with delayed weaning in the intensive care unit were completed through the joint efforts of medical, nursing and technical staff. The success rate of weaning was the main result, and the diaphragm mobility, diaphragm thickness and diaphragm thickening fraction in the diaphragm ultrasound results were the secondary results to conduct this study. The aim is to further clarify the impact of inspiratory muscle strength training on the successful weaning of patients with delayed weaning and the improvement of diaphragmatic function through clinical treatment and data collection and analysis.

In conclusion, IMT helps improve diaphragmatic function, and the improvement of diaphragmatic function will promote the improvement of respiratory function in patients, which also has certain clinical significance for accelerating weaning from the ventilator. Under the condition that our department is equipped with multiple physical therapists with experience in implementing IMT, the assessment and intervention of patients with delayed weaning in the intensive care unit were completed through the joint efforts of medical, nursing and technical staff. The success rate of weaning was the main result, and the diaphragm mobility, diaphragm thickness and diaphragm thickening fraction in the diaphragm ultrasound results were the secondary results to conduct this study. The aim is to further clarify the impact of inspiratory muscle strength training on the successful weaning of patients with delayed weaning and the improvement of diaphragmatic function through clinical treatment and data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received therapy in the HDU of the Respiratory Rehabilitation Center of Beijing Rehabilitation Hospital Affiliated to Capital Medical University and met the PMV criteria clearly recommended by the NAMDRC consensus in 2005, which is "mechanical ventilation for at least 6 hours a day for 21 consecutive days".

  * The patients' conditions were relatively stable, they were conscious, had no intellectual disability, no mental illness, no cognitive impairment, and gave informed consent.

    * They had spontaneous breathing and could tolerate short periods of being off the ventilator to complete the training.

      * The ventilator parameters met the following requirements: PEEP ≤ 10 cmH2O, FiO2 < 0.60, RR < 25.

Exclusion Criteria:

1) brain injuries, pulmonary contusions and lacerations, rib fractures, unhealed wounds in the chest and abdomen, etc. The condition is severe, and inspiratory muscle training and diaphragm ultrasound assessment cannot be performed. 2) No spontaneous breathing, completely dependent on mechanical ventilation; 3) Pre-existing pulmonary infection or severe heart, lung or kidney diseases before clinical trials, with unstable hemodynamics; 4) Poor cognitive function, poor compliance, and non-cooperation with treatment.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
weaning success rate | From enrollment to the end of treatment at 12 week

SECONDARY OUTCOMES:
Diaphragmatic function | from enrollment to the end of the treatment at 12 weeks
  DE in centimeter、thickness in millimeter、DTF in proportion
maximal inspiratory pressure | from enrollment to the end of the treatment at 8 weeks
EQ-5D-5L | From enrollment to the end of the intervention at 12 week
FVC(forced vital capacity) | from enrollment to the end of the ventilation at 12 week
  FVC in liters